CLINICAL TRIAL: NCT04101591
Title: Species Identification and Concentration Measurement of Antioxidants and Cytokines in the Anterior Chamber From Patients of Various Ocular Disorders
Brief Title: Identification and Measurement of Antioxidants and Cytokines in the Anterior Chamber of Various Ocular Disorders
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201900017B0
Record Dates: First submitted 2019-09-22; First posted 2019-09-24 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Eye Diseases
MeSH Terms: conditions — Eye Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Separated from the systemic circulation by a blood-aqueous barrier, the aqueous humor is secreted by the ciliary process (epithelium) of the ciliary body, and fills up the anterior and posterior chambers, with a total volume of 0.15 mL ~ 0.3mL. The major constituent if water (98.7％), with minimal amount chlorides, proteins, ascorbic acid, urea, and inorganic salts. The aqueous humor presents mild alkaline with a pH value of 7.3 ~ 7.5, while its specific gravity falls between 1.002 and 1.012. The functions of aqueous humor includes 1) to preserve the shape and integrity of the globe and to maintain the intraocular pressure within normal ranges; 2) to nourish the cornea, lens, and vitreous; 3) and to provide cellular or humoral immunity in case of intraocular inflammation or infection.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study offers evaluation and treatment for patients with corneal or retinal diseases, such as corneal opacities or diabetic retinopathy. The protocol is not designed to test new treatments; rather, patients will receive current standard of care treatments. The purpose of the study is twofold: 1) to allow ophthalmologist at Chang Gung Memorial Hospital (CGMH) to increase their knowledge of altered microenvironment in the corneal or retinal disorders and identify new pathways of possible research in this area; and 2) to establish a list of patients who may be qualified for new research as they are recruited. (Participants in this protocol will not be required to join a new study; the decision is dependent on the patients themselves.) Participants will be followed at least 3 months. Follow-up visits are scheduled according to the standard of care for the individual patient's ocular problems. Visual acuity and intraocular pressure will be checked at each visit, and some of the screening tests described above may be repeated to follow the progress of disease and evaluate the response to treatment.

DETAILED DESCRIPTION:
The primary purpose of the protocol is to accumulate a cohort of patients with corneal or retinal diseases for possible participation in new CGMH clinical trials and epidemiological protocols. Also, by providing long-term follow-up and treatment for a variety of corneal or retinal disorders, the relevant specialists and basic scientists at CGMH will be better able to identify research hypotheses about these diseases in addition to maintaining their clinical skills. The availability of cohorts of patients with a spectrum of corneal or retinal disorders will be valuable for the training of fellows in external eye or intraocular diseases, an important mission of the CGMH. The ability to provide long-term follow-up and care will also facilitate referral efforts for new CGMH protocols.

The corneal or retinal specialists at the Chang Gung Memorial Hospital will be free to choose those ocular disorders that interest them. However, the total number of patients that can be enrolled in the protocol will be restricted. This protocol is not designed to test any new treatments. Any evaluations or treatment under this protocol will be based on the current standard of care for each corneal or retinal diseases.

Participants in this patient evaluation and treatment protocol will be evaluated for potential eligibility in any new CGMH clinical trials or epidemiologic protocols as they are developed. If eligible, patients may be asked to participate in the new protocol. However, they will not be required to enter any protocol and their decision to participate will be entirely voluntary. No more than 200 patients will be accepted in this "Evaluation and Treatment Protocol."

ELIGIBILITY:
Inclusion Criteria:

* Intravitreal injection of patients
* Patients with vitreoretinal surgery
* Corneal transplant patients
* General cataract surgery patients

Exclusion Criteria:

* Those who have previously received aqueous extraction or intraocular surgery
* Eyeball infection patients
* Patients with uveitis
* Those with high intraocular pressure (>40 mmHg) or too low (<5 mmHg)

Ages: 1 Month to 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Subject inclusion criteria:
  1. No age limit
  2. Intravitreal injection of patients (such as: diabetic retinopathy, retinal vein occlusion, age-related macular degeneration Wait)
  3. Patients with vitreoretinal surgery (such as retinal detachment, macular wrinkles, macular holes, etc.), 4 corneal transplant patients (such as keratoconus, corneal opacity, corneal endothelial dystrophy, etc.)
  5. General cataract surgery patients
  Subject exclusion criteria:
  1. Eyeball infection patients (such as epidemic keratoconjunctivitis, corneal ulcer, endophthalmitis, etc.)
  2. Patients with uveitis (such as iridocyclitis, cytomegalovirus iriditis, toxoplasma retinal choroiditis, etc.)
  3. Those with high intraocular pressure (>40 mmHg) or too low (<5 mmHg)
  4. Those who have previously received aqueous extraction or intraocular surgery (such as cataract, vitrectomy, corneal transplantation, etc.)
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-01-16 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
The Correlation between the Total Antioxidative Capacity (TAC) and Ascorbic Acid (Vit C) | 5month
  Most of the antioxidant capacity of aqueous humor comes from vitamin C, and there is a positive correlation between the two.

CONTACTS AND LOCATIONS:
Overall Officials: Hung-Chi CHEN, PhD degree, Study Chair — Chang Gung Memorial Hospital
Locations (1):
- ChangGungMH, Taoyuan District, Taoyuan City, Taiwan

IPD SHARING:
Plan to Share IPD: No